CLINICAL TRIAL: NCT07293169
Title: H.Pylori Infection Among Women With Recurrent Abortion of Unknown Cause
Brief Title: Helicobacter Pylori Infection Among Women With Recurrent Abortion of Unknown Cause
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Gamal Ahmed Mostafa, Helicobacter pylori infection among women with recurrent abortion of unknown cause, Assiut University
Other Study IDs: H.pylori infection e abortion
Record Dates: First submitted 2025-11-22; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Helicobacter Pylori Infection, Susceptibility to

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group of women with history of recurrent abortion: another group of women without recurrent of abortion
  Interventions: Diagnostic Test: H pylori eradication

INTERVENTIONS:
Diagnostic Test: H pylori eradication — h.pylori stool antigen

SUMMARY:
* Helicobacter pylori (H. pylori) infection affects approximately one half of the world population and it is more prevalent in developing countries. This microorganism colonizes the stomach. Typically, it is acquired during childhood and causes asymptomatic chronic infection. A small portion of H. pylori infected subjects develop peptic ulcers and gastric carcinoma, usually during late adulthood. (1,2)
* Some studies show a relationship between H.pylori and pregnancy-related disorders, such as fetal growth defects and malformations, miscarriage and, more recently, to pre-eclampsia. (3)
* Abortion is one of the most common complications of pregnancy. Infection is one of the main causes of abortion, a cause which is more important in spontaneous abortion; infections account for only 5% of recurrent abortions. (4)
* The severity of infection with H.pylori: given the increasing secretion of inflammatory cytokines and CD8 +, CD4 + in T cells and increasing interferons (IFN), studies have shown that infection with Helicobacter pylori activates immune cells in the uterus and endometrial surface cells, increases TH1 response to helicobacter, disturbs the ratio of T-Helper 2 / T-Helper 1 cytokines, causes abnormalities in the formation of natural vessels in the uterus and, ultimately, leads to abortion.(5)
* Repeated spontaneous abortion (RSA): >=2 consecutive spontaneous pregnancy losses before 20 weeks gestation.(6)
* To determine if H.pylori infection is significantly associated with recurrent abortion of unknown cause........

DETAILED DESCRIPTION:
3.Patients and methods

Study design:

Case Control study two groups (one group of 50 women with history of recurrent abortion and another group of 50 women without recurrent of abortion)

Study location:

the study will be conducted in Assiut university hospitals (women's health hospital) .

Study duration:

the study will be carried out from October 2025 till October 2026.

Sample size :

the calculated sample size for two groups 100 cases (one group of 50 women with history of recurrent abortion and another group of 50 women without recurrent of abortion).

4.Inclusion criteria

* All woman with repeated abortion of Unknwon cause.
* Not received H.pylori eradication therapy in prior 3 months .

  5.Exclusion criteria
* Known uterine anatomical causes of abortion.
* Current systemic antibiotic use and PPIs within 2 weeks.
* Medical diseases as (Thyroid disorders , DM,HTN).
* Antiphspholipid syndrome. 6.Methods
* Case Control study at Assiut woman's heath hospital from October 2025 till October 2026.
* Case Control study two groups (one group of women with history of recurrent abortion and another group of women without recurrent of abortion) by stool antigen test.

  7.All patients will be subjected to the following
* Complete obstetric history , medical history, smoking ,alcohol, recent antibiotics ,PPIs , socioeconomic status
* Laboratory samples :

H.pylori antigen in stool ,complete blood count , abdominopelvic ultrasound , urine analysis , liver and kidney function tests ,TSH , prolactin and any necessary investigation will be done.

Anti cardiolipin (IgM , IgG) ,Lupus anti coagulant and Anti B2 glycoproteinA1 (IgM, IgG) and 3D US on uterus . 8.Ethical considerations

* All subjects will provide written informed consent to participate in the study .
* The protocol of the study will be presented to the local ethics committee for approval.

  9.Statistical analysis
* Statistical analysis will be performed using Spss version 23.

  10.References
* 1. Malaty HM. Epidemiology of Helicobacter pylori infection. Best Pract Res Clin Gastroenterol 2007; 21: 205-214
* 2. Suerbaum S, Michetti P. Helicobacter pylori infection. N Engl J Med 2002; 347: 1175-1186
* 3. Chen MJ, Fang YJ, Wu MS, Chen CC, Chen YN, Yu CC et al. Application of Helicobacter pylori stool antigen test to survey the updated prevalence of Helicobacter pylori infection in Taiwan. 2020;35:233-40
* 4. Ambühl LM, Baandrup U, Dybkær K,Blaakær J, Uldbjerg N, Sørensen S. Human papillomavirus infection as a possible cause of spontaneous abortion and spontaneous preterm delivery 2016;2016.
* 5. Azami M, Nasirkandy MP, Mansouri A, Darvishi Z, Rahmati S, Abangah G, DehghanHR, Borji M, Abbasalizadeh S. GGollobal Prevelance of H.pylori infection in pregnant women: a systematic review and meta-analysis study. Int J Women's Health Reprod Sci. 2017;5:30-6.
* 6. Practice Committee of the American Society for Reproductive Medicine. Definitions of infertility and recurrent pregnancy loss: a committee opinion. Fertil Steril. 2013 99:63.

ELIGIBILITY:
Inclusion Criteria• All woman with repeated abortion of Unknwon cause.

* Not received H.pylori eradication therapy in prior 3 months .

Exclusion Criteria:

* Known uterine anatomical causes of abortion.
* Current systemic antibiotic use and PPIs within 2 weeks.
* Medical diseases as (Thyroid disorders , DM,HTN).
* Antiphspholipid syndrome.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — * All woman with repeated abortion of Unknwon cause.
  * Not received H.pylori eradication therapy in prior 3 months .
Study Population: • All woman with repeated abortion of Unknwon cause.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
• To determine if H.pylori infection is significantly associated with recurrent abortion of unknown cause | baseline
H.pylori infection among women with recurrent abortion of unknown cause | the study will be carried out from October 2025 till October 2026
  • To determine if H.pylori infection is significantly associated with recurrent abortion of unknown cause........